CLINICAL TRIAL: NCT00283400
Title: Treatment of Subarachnoid Hemorrhage With Human Albumin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study met safety endpoints
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jose I. Suarez, Professor of Neurology, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01NS049135 (NIH); R01NS049135 (NIH)
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Subarachnoid Hemorrhage
Keywords: subarachnoid hemorrhage; SAH; human albumin; HA; cerebral vasospasm; aneurysm; neuroprotective
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Aneurysm | interventions — Serum Albumin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- dosage tier 1 (Active Comparator): 0.625 g/kg 25% human albumin
  Interventions: Drug: 25% human albumin
- dosage tier 2 (Active Comparator): 1.25 g/kg 25% human albumin
  Interventions: Drug: 25% human albumin
- dosage tier 3 (Active Comparator): 1.875 g/kg 25% human albumin
  Interventions: Drug: 25% human albumin
- dosage tier 4 (Active Comparator): 2.5 g/kg 25% human albumin
  Interventions: Drug: 25% human albumin

INTERVENTIONS:
Drug: 25% human albumin — 25% human albumin: after approval by the Data and Safety Monitoring Board dosage tier would be escalated to the subsequent higher level sequentially.

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of 25 percent human albumin therapy in patients with subarachnoid hemorrhage.

DETAILED DESCRIPTION:
An estimated 37,500 people in the United States have subarachnoid hemorrhage (SAH) every year. SAH is usually secondary to a brain aneurysm that has burst. In SAH the bleeding accumulates around the lining of the brain. SAH is associated with a 51percent mortality rate, and one third of survivors are left functionally dependent. Cerebral vasospasm, which is a delayed narrowing of the cerebral arteries following SAH, has been identified as the most important reason for neurological deterioration and bad outcome in cases of SAH. Cerebral vasospasm may be caused by multiple mechanisms.

Treatment with a neuroprotective agent, such as human albumin (HA), may be beneficial for prevention of cerebral vasospasm and improved clinical outcome in patients with SAH. HA is a major protein found in blood and is responsible for maintaining fluid balance in the vascular system (blood vessels). The purpose of this study was to determine the safety and tolerability of 25 percent HA therapy in patients with SAH. This open-label, dose-escalation study will provide necessary information for a future definitive phase III clinical trial on the efficacy of treatment with HA in patients with SAH.

The study was designed to enroll 80 patients at 5 centers in the US. Patients with eligible SAH first underwent surgical or endovascular repair, which was considered standard care. Endovascular repair was a repair of the aneurysm from the inside of the blood vessel.

Following neurosurgical or endovascular treatment, participants were given a daily infusion of HA for 7 days. The HA dose was allocated as follows: the first tier (20 patients) would receive 0.625 grams (g) of HA per kilogram (kg) of body weight; patients in the second tier would receive 1.25g of HA per kg; patients in the third tier would receive 1.875g of HA per kg; and patients in the fourth tier would receive 2.5g of HA per kg. Safety and tolerability was evaluated by the Data and Safety Monitoring Board (DSMB) after each tier was completed and before the study advanced to the next dose tier. A specific safety threshold for congestive heart failure and other adverse events was defined based on data from previous studies.

In the follow-up phase, patients participated in study-related evaluations of their health at 15 days and three months. Duration of the study for participants was 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) were at least 18 but younger than 80 years of age.
* Onset of new neurological signs of subarachnoid hemorrhage within 72 hours at the time of evaluation and initiation of treatment with 25% human albumin.
* Clinical signs consistent with the diagnosis of subarachnoid hemorrhage including severe thunderclap headache, cranial nerve abnormalities, decreased level of consciousness, meningismus and focal neurological deficits.
* Computed tomography demonstrated subarachnoid hemorrhage.
* Cerebral angiography revealed the presence of saccular aneurysm(s) in a location that explains the subarachnoid hemorrhage.
* Treatment of cerebral aneurysm was carried out prior to initiation of HA infusion but within 72 hours of symptom onset. Accepted treatments of aneurysms include surgical clipping or endovascular embolization.

Exclusion Criteria:

* Time of symptom onset could be reliably assessed.
* No demonstrable aneurysm by cerebral angiography.
* Evidence of traumatic, mycotic, or fusiform aneurysm by cerebral angiography.
* World Federation of Neurological Surgeons scale of IV and V
* Computed tomography scale of 0-1
* History within the past 6 months, and/or physical findings on admission of decompensated congestive heart failure (NYHA Class IV or congestive heart failure requiring hospitalization).
* Patient received albumin prior to treatment assignment during the present admission.
* Hospitalization for or diagnosis of acute myocardial infarction within the preceding 3 months.
* Symptoms or electrocardiographic signs indicative of acute myocardial infarction on admission.
* Electrocardiographic evidence and/or physical findings compatible with second- or third-degree heart block, or of cardiac arrhythmia associated with hemodynamic instability.
* Echocardiogram performed before treatment revealing a left ventricular ejection fraction ≤ 40% (if available).
* Serum creatinine > 2.0 mg/dl or creatinine clearance < 50 ml/min.
* Pregnancy, lactation or parturition within previous 30 days.
* Allergy to albumin.
* Severe prior physical disability that precludes evaluation of clinical outcome measures.
* History of chronic lung disease
* Current participation in another drug treatment protocol.
* Severe terminal disease with life expectancy less than 6 months.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-01; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose I. Suarez, MD, Principal Investigator — Baylor College of Medicine
Locations (6):
- United States (4):
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Penn State University, Hershey, Pennsylvania
  - Data Coordination Unit, Department of Biostatistics, Bioinformatics and Epidemiology, at the Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Toronto, Toronto, Ontario

REFERENCES:
- [Background] Suarez JI, Shannon L, Zaidat OO, Suri MF, Singh G, Lynch G, Selman WR. Effect of human albumin administration on clinical outcome and hospital cost in patients with subarachnoid hemorrhage. J Neurosurg. 2004 Apr;100(4):585-90. doi: 10.3171/jns.2004.100.4.0585. PMID 15070109
- [Background] Suarez JI, Qureshi AI, Yahia AB, Parekh PD, Tamargo RJ, Williams MA, Ulatowski JA, Hanley DF, Razumovsky AY. Symptomatic vasospasm diagnosis after subarachnoid hemorrhage: evaluation of transcranial Doppler ultrasound and cerebral angiography as related to compromised vascular distribution. Crit Care Med. 2002 Jun;30(6):1348-55. doi: 10.1097/00003246-200206000-00035. PMID 12072693
- [Background] Lennihan L, Mayer SA, Fink ME, Beckford A, Paik MC, Zhang H, Wu YC, Klebanoff LM, Raps EC, Solomon RA. Effect of hypervolemic therapy on cerebral blood flow after subarachnoid hemorrhage : a randomized controlled trial. Stroke. 2000 Feb;31(2):383-91. doi: 10.1161/01.str.31.2.383. PMID 10657410
- [Background] Haley EC Jr, Kassell NF, Torner JC. A randomized controlled trial of high-dose intravenous nicardipine in aneurysmal subarachnoid hemorrhage. A report of the Cooperative Aneurysm Study. J Neurosurg. 1993 Apr;78(4):537-47. doi: 10.3171/jns.1993.78.4.0537. PMID 8450326
- [Background] Wilkes MM, Navickis RJ. Patient survival after human albumin administration. A meta-analysis of randomized, controlled trials. Ann Intern Med. 2001 Aug 7;135(3):149-64. doi: 10.7326/0003-4819-135-3-200108070-00007. PMID 11487482
- [Background] Finfer S, Bellomo R, Boyce N, French J, Myburgh J, Norton R; SAFE Study Investigators. A comparison of albumin and saline for fluid resuscitation in the intensive care unit. N Engl J Med. 2004 May 27;350(22):2247-56. doi: 10.1056/NEJMoa040232. PMID 15163774
- [Background] Belayev L, Liu Y, Zhao W, Busto R, Ginsberg MD. Human albumin therapy of acute ischemic stroke: marked neuroprotective efficacy at moderate doses and with a broad therapeutic window. Stroke. 2001 Feb;32(2):553-60. doi: 10.1161/01.str.32.2.553. PMID 11157196
- [Background] Osterloh K, Ewert U, Pries AR. Interaction of albumin with the endothelial cell surface. Am J Physiol Heart Circ Physiol. 2002 Jul;283(1):H398-405. doi: 10.1152/ajpheart.00558.2001. PMID 12063314
- [Background] Zhang WJ, Frei B. Albumin selectively inhibits TNF alpha-induced expression of vascular cell adhesion molecule-1 in human aortic endothelial cells. Cardiovasc Res. 2002 Sep;55(4):820-9. doi: 10.1016/s0008-6363(02)00492-3. PMID 12176131
- [Result] Suarez JI, Martin RH, Calvillo E, Dillon C, Bershad EM, Macdonald RL, Wong J, Harbaugh R; ALISAH Investigators. The Albumin in Subarachnoid Hemorrhage (ALISAH) multicenter pilot clinical trial: safety and neurologic outcomes. Stroke. 2012 Mar;43(3):683-90. doi: 10.1161/STROKEAHA.111.633958. Epub 2012 Jan 19. PMID 22267829
- [Result] Suarez JI, Martin RH, Calvillo E, Bershad EM, Venkatasubba Rao CP. Effect of human albumin on TCD vasospasm, DCI, and cerebral infarction in subarachnoid hemorrhage: the ALISAH study. Acta Neurochir Suppl. 2015;120:287-90. doi: 10.1007/978-3-319-04981-6_48. PMID 25366638

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The National Institutes of Health funded the Albumin in Subarachnoid Hemorrhage (ALISAH) pilot study, initiated in May 2006 and terminated in May 2010. The study was originally planned for 3 years but mostly due to the principal investigators transferring institutions and initiation of 2 non-US sites, 1 extra year was needed.
Groups:
- Dosage Tier 1: 25% human albumin 0.625 g/kg
- Dosage Tier 2: 25% human albumin 1.25 g/kg
- Dosage Tier 3: 25% human albumin 1.875 g/kg
- Dosage Tier 4: 25% human albumin2.5 g/kg
Period: Overall Study
Arm/Group | Dosage Tier 1 | Dosage Tier 2 | Dosage Tier 3 | Dosage Tier 4
Started | 20 | 20 | 7 | 0
Completed | 18 | 19 | 6 | 0
Not Completed | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dosage Tier 4: 25% human albumin 2.5 g/kg
- Total: Total of all reporting groups
Arm/Group | Dosage Tier 1 | Dosage Tier 2 | Dosage Tier 3 | Dosage Tier 4 | Total
Number analyzed (Participants) | 20 | 20 | 7 | 0 | 47
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 | 0 |  | 0
  Between 18 and 65 years | 19 | 19 | 6 |  | 44
  >=65 years | 1 | 1 | 1 |  | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (25) | 51 (24) | 55 (25) |  | 51 (25)
Gender [Number; unit: participants]
  Female | 15 | 13 | 6 |  | 34
  Male | 5 | 7 | 1 |  | 13
Region of Enrollment [Number; unit: participants]
  United States | 15 | 12 | 4 |  | 31
  Canada | 5 | 8 | 3 |  | 16

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of the 25% Human Albumin Dosages and the Functional Outcome.
Description: Tolerability outcome: Subject's ability to receive the full allocated human albumin dose without incurring frank congestive heart failure or experiencing anaphylactic reactions that required discontinuation of the treatment. Study would be terminated if 2 or more subjects developed severe or life-threatening heart failure considered to be related (probably, possibly, and definitely) to albumin treatment.
Time Frame: 9 days after enrollment
Population: Sample size consideration for this Phase I dose-escalation study was based on the feasibility of recruiting patients in a 3-year study period at 5 sites.The recruitment yield would be a maximum of 80 patients or 20 patients per dosage group. Statistical analyses were mainly descriptive.
Measure: Number; unit: participants
Arm/Group | Dosage Tier 1 | Dosage Tier 2 | Dosage Tier 3 | Dosage Tier 4
Number analyzed (Participants) | 20 | 20 | 7 | 0
participants | 0 | 1 | 2 |

2. Secondary Outcome: Serious Adverse Events
Description: Serious adverse events included neurological and medical complications and neurological deterioration.
  Neurological deterioration was defined as a decline by more than 2 points in the Glasgow Coma Scale.
Time Frame: within 3 months after enrollment
Measure: Number; unit: participants
Arm/Group | Dosage Tier 1 | Dosage Tier 2 | Dosage Tier 3 | Dosage Tier 4
Number analyzed (Participants) | 20 | 20 | 7 | 0
participants
  Symptomatic Cerebral Vasospasm | 4 | 3 | 2 |
  Pulmonary Edema | 2 | 2 | 0 |
  ARDS | 0 | 0 | 1 |
  Rebleeding | 1 | 0 | 0 |
  Pulmonary Embolism | 1 | 0 | 0 |
  Gram-Negative Ventriculitis | 1 | 0 | 0 |
  Hypotension due to sepsis | 1 | 0 | 0 |

3. Secondary Outcome: Good Clinical Outcome Was Defined as a Glasgow Outcome Scale Score of 0-1
Description: Number of subjects with good clinical outcome defined as a Glasgw Outcome Scale score of 0-1
Time Frame: 3 months after enrollment
Measure: Number; unit: participants
Arm/Group | Dosage Tier 1 | Dosage Tier 2 | Dosage Tier 3 | Dosage Tier 4
Number analyzed (Participants) | 20 | 20 | 7 | 0
participants | 13 | 17 | 3 |
Statistical Analysis 1: Comparison: Dosage Tier 1 vs Dosage Tier 2; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Post-hoc comparison of outcomes in dosage tier 1 vs dosage tier 2; Odds Ratio (OR) = 3.05, 95% CI 2-sided [0.65 to 14.1]

ADVERSE EVENTS:
Arm/Group | Dosage Tier 1 | Dosage Tier 2 | Dosage Tier 3 | Dosage Tier 4
Serious Adverse Events (participants affected / at risk) | 5/20 | 3/20 | 3/7 | 0/0
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/7 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dosage Tier 1 (N=20) | Dosage Tier 2 (N=20) | Dosage Tier 3 (N=7) | Dosage Tier 4 (N=0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Severe or life-threatening acute heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Symptomatic Cerebral Vasospasm (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2) | 0 (0)
Rebleeding (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gram-negative ventriculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hypotension due to sepsis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Our study has several limitations. ALISAH is an early phase design and we do not have concurrent controls. In addition, the study was neither randomized nor powered to test for efficacy effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No